CLINICAL TRIAL: NCT01419405
Title: Pregabalin Has Additive Analgesic and Ventilatory Depressive Effects in Combination With Remifentanil
Brief Title: Pregabalin and Remifentanil - Analgesia and Ventilation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011/1380-1
Record Dates: First submitted 2011-06-30; First posted 2011-08-18 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Pain
Keywords: analgesia; acute experimental pain; cold pressor test; pregabalin; remifentanil
MeSH Terms: conditions — Pain; Agnosia | interventions — Pregabalin; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pregabalin/placebo (Experimental)
  Interventions: Drug: Pregabalin
- placebo/remifentanil (Active Comparator)
  Interventions: Drug: Remifentanil
- placebo/placebo (Placebo Comparator)
  Interventions: Drug: sugar pill, saline infusion
- Pregabalin/Remifentanil (Experimental)
  Interventions: Drug: Pregabalin; Drug: Remifentanil

INTERVENTIONS:
Drug: Pregabalin — hard capsule, 150 mg, 2 times, 2 days
  Other Names: Lyrica
  Arms: Pregabalin/Remifentanil; Pregabalin/placebo
Drug: Remifentanil — 50-90 min: TCI 0.6 ng/mL, 100-140 min: 1.2 ng/mL, 150-190 min: TCI 2.4 ng/mL
  Other Names: Ultiva
  Arms: Pregabalin/Remifentanil; placebo/remifentanil
Drug: sugar pill, saline infusion — hard capsule, 150 mg, 2 times, 2 days, saline infusion
  Other Names: Laktose monohydrat; NaCl 0,9%
  Arms: placebo/placebo

SUMMARY:
In this experimental study on healthy volunteers we explored the effect of pregabalin alone and in combination with remifentanil on acute experimental pain and ventilatory function.

DETAILED DESCRIPTION:
Pain during cold pressor test (CPT) was scored at all dose levels of remifentanil on a visual analogue scale (VAS 0-100 mm). Ventilatory function was measured by spirometry registering respiratory frequency (breaths/min), minute volume (L/min) and expiratory end-tidal carbon dioxide tension (mmHg).

Side effects such as nausea and sedation were registered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers,
* > 18 yrs < 55 yrs,
* negative pregnancy test

Exclusion Criteria:

* Pregnancy,
* nursing,
* known heart-, lung- or liver disease,
* kidney failure/peptic ulcers,
* use of liver enzyme-inducing medications,
* known allergy against the medications used in the trial,
* use of psychotropic drugs, analgesics or alcohol used the last 24 hours before the trial,
* body weight > 100 kg or 30% deviation from normal weight,
* participant in other studies during the last 2 months,
* individuals who do not master Norwegian language

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 123 sec x 4
  Pain was caused by Cold Pressure Test

SECONDARY OUTCOMES:
Ventilatory function | 10 min x 4
  Respiratory frequence (breath/min), tidal volume (mL), minute volume (L)and expiratory end-tidal carbon dioxide tension (mmHg)
Cognitive function | 4 min x 4
  Cognitive function was tested using pc-tests like Cambridge Neuropsychological Test Automated Battery (CANTAB) and Stroop-test

CONTACTS AND LOCATIONS:
Overall Officials: Audun Stubhaug, MD, DMedSci, Prof., Principal Investigator — Oslo University Hospital HF, Division of Critical Care
Locations (1):
- Oslo Universitetssykehus, Rikshospitalet, Oslo, Norway